CLINICAL TRIAL: NCT01518010
Title: Multi-player Online Video Games for Cognitive Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Portsmouth (Other)
Responsible Party: Principal Investigator, Jason Colman, Principal Investigator, University of Portsmouth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: COLMAN
Record Dates: First submitted 2012-01-15; First posted 2012-01-25 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Acquired Brain Injury
Keywords: Brain injury; Cognitive rehabilitation; Video game
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GamePlay (Experimental)
  Interventions: Behavioral: Play game

INTERVENTIONS:
Behavioral: Play game — Participants engage in non-game activity (establish baseline) 7 * 1 hr weekly; play single-player game 7 * 1 hr weekly; play multi-player game 7 * 1 hr weekly.

SUMMARY:
This research project aims to find out if a multiplayer online video game can provide therapeutic benefit for people who have survived a brain injury.

Video games provide therapeutic benefits in many contexts (Griffiths, 2005). Players of online multiplayer games behave altruistically and form friendships (Wang and Wang, 2008). These positive emotional effects may enhance cognitive rehabilitation, because the cognitive and emotional sides of rehabilitation are connected (Mateer, 2005).

The hypothesis is thus: that playing multiplayer online games can be a useful form of cognitive rehabilitation for brain-injured people.

This research will identify whether or not multi-player online video games may be used as a complementary therapeutic tool. A further aim is to develop guidelines which would help others considering the use of video games for cognitive rehabilitation.

DETAILED DESCRIPTION:
Purpose and design

This research aims to find out if massively multi-player online games (MMOs), a relatively new type of video game, can be used as a form of therapy for people who have survived an acquired brain injury.

Numerous previous studies have shown that video games can be used as therapy in many contexts. However, there is some evidence that video games are not an effective form of cognitive rehabilitation for brain injury survivors (Malec et al., 1984). The difference in this research is that MMOs incorporate social interaction into the game play experience. It is proposed that this strengthening of social bonds will be more beneficial than a similar single-player game.

Due to the narrow focus of the research it is anticipated that the number of potential participants will be small, on the order of ten participants. It is recognised that such a small sample size is not compatible with a randomised controlled trial. Instead, the research will employ a single-subject research design, where a higher number of participants will strengthen the external validity of the results.

The research question and design have been developed primarily by the Chief Investigator (PhD student), with critique from the supervisory team. Feedback has also been received from healthcare professionals who have been contacted by the C.I.

Participants will be asked for their feedback on a video game and its user interface. This is to ensure that the video game is suitable for the participant, and that the participant is able to play it. This stage is expected to consist of three or four sessions of 30 mins duration, every 2 weeks.

Participants will then be asked to play the video game for a number of sessions. The number of sessions is 21. The duration of each session is one hour. The sessions are to be held once per week.

Null/alternative hypotheses

The null hypotheses are that a single-player video game will not improve cognitive skills; and that a multi-player online video game will not improve cognitive skills. The alternative hypotheses are that a single-player game will improve cognitive skills, and a multi-player online game will provide further improvement.

Study design

The first stage of the research will be to design and refine a prototype online multi-player video game, working in collaboration with participants, firstly able-bodied, and then disabled. The researcher will work with each participant to develop a user interface which enables him or her to play the video game.

The study will then employ a single-case research design for each disabled participant. An RCT would not be valid given the expected number of participants. Time-series data will be collected in three phases: to obtain a baseline; to measure the effects of a single-player video game; and to measure the effects of a multi-player online game. Each phase has seven sessions. The sessions are one hour, weekly.

During the baseline phase, The participant will engage in a non-game task using the interface defined in the pre-trial phase. This phase may compensate for researcher effects. For the next phase, the participant will engage in a single-player version of the video game. For the final phase, the participant will engage in a multi-player online game.

Player activity in the single- and multi-player games will be logged for analysis. Interviews with participants will be used to build a thick narrative of each participants' experience over the course of the study.

Recruitment

Participants will be recruited by contacting head injury units, day care centres, and organisations such as Headway and the ARNI Trust. The C.I. will meet with potential participants who express an interest in the study.

A cornerstone of rehabilitation is that the goals are relevant to the client's everyday life. Therefore the details of how any individual's cognitive improvements will be measured must be based on a dialogue with each individual.

Consent

Informed consent must be given by a participant before any involvement in the study.

A participant information sheet will be provided. The C.I. will be present to talk through the issues with the participant. The NHS guidelines for writing clear information sheets will be followed.

Due to the nature of the participants' injuries, particular care and emphasis is placed on establishing capacity to give consent. The Department of Health gives guidelines on gauging capacity but family members and care workers will be a key source of guidance.

It is expected that participants will provide a written signature on a consent form, but again due to the nature of the participant's injuries this may not be possible. In this case the verbal consent of the participant would be recorded and witness(es) would sign the form.

Risks, burdens and benefits

The main medical risk of playing video games is the possibility of epileptic seizure due to photosensitive epilepsy, (PSE). Minor risks are: the possibility of aches and pains; eye strain; and stress caused by extended periods of vigilance. These risks are mitigated by conducting the research at day care centres where medical staff will be on hand, and by limiting play to one hour per week, broken into smaller play sessions (e.g. 3 * 20 mins). Additionally, again to minimise risk of photosensitive seizure, screen luminance will be kept to a minimum.

Other issues to consider when using video games as therapy are: video game "addiction"; violent content; and the offensive nature of some games. The issue of any potential addiction is mitigated by the short playing times; the issue of game suitability will be managed by previewing and discussing game content with participant, family members and carers as appropriate.

Potential benefits to participants: Playing a suitable game should provide feelings of well-being and improved self esteem. With the added social aspect of multi-player online games, participants could also feel less isolated. These improvements in emotional health may have beneficial effects on cognitive skills such as communication.

Confidentiality

Participant personal details will be kept confidential. When data is reported, random numeric IDs will be used to refer to individuals. Guidelines issued by the Office of National Statistics will be followed when tabulated data contains cells with zeros or extremely low numbers, so that potential identification of participants is prevented.

ELIGIBILITY:
Inclusion Criteria:

* Have survived an acquired brain injury
* Have progressed through the acute stage of treatment and rehabilitation
* Be attending a day centre periodically
* Have an interest in playing video games
* Be physically capable of playing a video game, with adjustments to the user interface as required
* Be capable of giving or withholding consent
* Have access to suitable computer with internet access at day centre

Exclusion Criteria:

* Any history of photosensitive epilepsy
* Any history of ill effects due to playing video games, or if any ill-effects are shown when playing video games
* On advice of medical staff or carer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Player in-game activity data | Time series data collected each hourly session, weekly, for 21 weeks
  All player activity is logged on server with timestamp. Data to be logged:
  * Player movement (ID, location, timestamp)
  * Messages sent (Sender and recipient IDs, text, timestamp)
  * In-game objects created or modified (participant ID, object ID, object type, timestamp)
  Each weekly session will produce one block of this data. The 21 blocks constitute time series data which will be analysed for evidence of improvement in cognitive skills.

SECONDARY OUTCOMES:
Player attitudes | Weekly , for 21 weeks
  Each session in debriefing, players will be asked about their attitudes and feelings about the effects of playing video games

CONTACTS AND LOCATIONS:
Overall Officials: Jason E Colman, Principal Investigator — University of Portsmouth

REFERENCES:
- [Background] Mateer, C. (2005) Fundamentals of cognitive rehabilitation. In Halligan, P., and Wade, D. (Eds.) Effectiveness of rehabilitation for cognitive defects. Oxford University Press
- [Background] Griffiths M. Video games and health. BMJ. 2005 Jul 16;331(7509):122-3. doi: 10.1136/bmj.331.7509.122. No abstract available. PMID 16020833
- [Background] Wang CC, Wang CH. Helping others in online games: prosocial behavior in cyberspace. Cyberpsychol Behav. 2008 Jun;11(3):344-6. doi: 10.1089/cpb.2007.0045. PMID 18537505
- [Background] Malec, J., Jones, R., Rao, N., Stubbs, K. (1984) Video game practice effects on sustained attention in patients with craniocerebral trauma. Cognitive Rehabilitation 2 (4): 18 - 23